CLINICAL TRIAL: NCT05178108
Title: Transposition of Dynamic MRI Data From Healthy Patients to an in Vitro Swallowing Simulator
Brief Title: Transposition of Dynamic MRI Data From Healthy Subjects to an in Vitro Swallowing Simulator
Acronym: SWALL-E
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 8260
Record Dates: First submitted 2021-10-22; First posted 2022-01-05 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Imaging Data Collection From Dynamic Swallowing MRI in Healthy Volunteers; Create Operating Algorithms; Apply the Imaging Data of MRI to a Swallowing Simulator
Keywords: dysphagia; deglutition in normal subjects; swallowing; robotic in-vitro simulation
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy individuals (Other)
  Interventions: Other: Real-time MRI of swallowing

INTERVENTIONS:
Other: Real-time MRI of swallowing — The examination recording a total of 9 sequences of less than 30 seconds will be performed, in transverse section (passing through the epiglottis), frontal section, in the plane of the posterior pharyngeal wall, and in median sagittal section.
  Each bolus of 20 ml will be administered in full, in one go, using a syringe. It is kept in the mouth for a few seconds and swallowed on demand.
  The semi-liquid bolus of 20 ml comes from the mixture of 198 ml of pineapple juice to 10 gr of Nutilis Powder (NUTRICIA), food thickener containing neither gluten, nor lactose.
  Ingredients: Dextrin-maltose, thickeners (modified starch (corn), tara gum, xanthan gum, guar gum).
  * 3 sequences with no food
  * 3 sequences with ingestion of a liquid bolus of 20 ml (pineapple juice) mouth closed
  * 3 sequences with ingestion of a semi-liquid bolus of 20 ml (pineapple juice + Nutilis Powder) mouth closed

SUMMARY:
Swallowing is a complex process, involving a very fine synchronization of the pharyngo-larynx, with respiration, under the control of the central nervous system and numerous peripheral effectors. Any dysfunction can lead to aspiration a source of morbidity and mortality.

These dysfunctions of the aerodigestive tract affect a considerable number of patients with multiple etiologies: squamous cell carcinoma of the upper aerodigestive tract, peripheral or central neurological dysfunctions, neurosurgical or neurovascular causes, geriatric pathologies and intensive care complications.

Aspiration pneumopathy is the most severe complication, which can lead to death. For decades, only techniques such as tracheotomy or enteral feeding (nasogastric tube/gastrostomy tube), associated or not with speech therapy, have been proposed to counter this problem. These invasive treatments remain symptomatic. These treatments bypass the pharyngolaryngeal dysfunction without resolving it and still significantly alter the patients' quality of life.

In 2012, a first worldwide clinical study (published in the NEJM) based on 6 patients, conducted by the ENT team in Strasbourg, demonstrated an improvement in the quality of life of patients who had undergone total laryngectomy, by proposing the placement of a titanium laryngeal implant equipped with an upper valve. This strategy intended to avoid aspiration of food hile allowing normal breathing. Although this technique did not solve all problems (the persistence of food going the wrong way), this study allowed a conceptual change in the attempt to solve swallowing problems by the introduction of pharyngolaryngeal implants.

The latter remains a challenge, but clinical trials of implants with a functional valve effected after removal of the larynx or on an existing but dysfunctional larynx have demonstrated the indivisibility of the pharynx-larynx couple in the search for permanent solutions.

This physiological process can be studied with imaging. Videofluoroscopy is the reference method allowing a dynamic study of swallowing. However, it does not allow the study of soft tissue movement and exposes the patient to repeated irradiation. Recently, MRI has shown its ability to visualize the entire pharyngolaryngeal structures accurately and dynamically during the swallowing process.

To improve the understanding and resolution of swallowing disorders, a unique robotic platform, consisting of a dynamic silicone skeleton reproducing the complexity of the pharyngolarynx, was initially developed by PROTIP MEDICAL (SWALL-E). This is the object of a French patent, transferred to the HUS University Hospitals of Strasbourg.

The aim this study is to correlate and calibrate this platform with dynamic MRI data in healthy subjects, by studying the movement of the different anatomical structures of the pharyngolarynx during swallowing movements (speed, amplitude and synchronization of the pharyngolarynx movements).

The immediate application of SWALL-E, after calibration and validation, will: i) allow the reproduction of a physiological swallowing mechanism; ii) allow to produce a pathological and personalized simulation of swallowing disorders in vitro; iii) allow the design of implants produced by 3D printing, and to analyze their effectiveness before implantation; iv) to modify in parallel and if necessary the rheology of the food boluses, thus contributing to a significant global improvement for the patient.

Thus, this platform, unique in its conception, aims not only at making a diagnosis of the specific pathology of the patient, but also aims at a personalized management adapted to the patient, inexistent until now.

Indeed, if the diagnostic methods are numerous (nasofibroscopy, swallowing transit, videofluoroscopy, study of swallowing noises by acoustic signals, swallowing cinetigraphy...), the treatments have remained identical for decades (speech therapy), and are not targeted (pharyngeal stimulation), despite the fact that each patient presents a specific pathology that is difficult to reunify under a "universal" treatment.

DETAILED DESCRIPTION:
To date, in vitro models of the pharyngeal phase of swallowing have led to limited results. No high-fidelity robot of the pharyngo-larynx has been developed.

For this purpose, a robotic device, called SWALL-E (21) was created. It is based on a realistic anatomical model of a human pharyngolaryngeal tract in which the anatomical structures and mechanisms involved in the pharyngeal swallowing phase are precisely actuated and controlled. It allows to simulate a swallow in terms of dynamics, size, and timing by reproducing the anatomical structures directly involved in the bolus transport process of the pharyngeal phase (tongue base retraction; vocal cords opening/closing; larynx elevation; pharynx contraction; epiglottis tilt; upper esophageal sphincter opening/closing). SWALL-E, illustrated below, was designed with the main goal of reproducing with maximum fidelity the anatomy and physiology of the pharyngeal phase of adult human swallowing The SWALL-E platform is currently operational but has not yet been calibrated.

The specifications were defined as follows: i) full-scale model of the adult human anatomical tract in a flexible material; ii) reproduction of the anatomical structures directly involved in the bolus transport process of the pharyngeal phase; iii) reproduction of the critical physiological mechanisms in an accurate and spatially and temporally adjustable manner.

The mechanisms reproduced are i) bolus injection; ii) tongue base retraction; iii) vocal cord opening/closing; iv) laryngeal elevation; v) pharyngeal contraction; vi) epiglottis tilt; vii) upper esophageal sphincter opening/closing.

The normal swallowing sequences performed demonstrated the ability of the system to reproduce the chronological order of biomechanical movements. This was achieved from clinical observations, and then adapted into a model whereby the movement and path of the food bolus can be physically imitated and controlled.

SWALL-E is thus able to simulate the in vitro pharyngolaryngeal phase of "normal" swallowing by achieving a transit time comparable to that found in a healthy subject without any misdirection.

The current SWALL-E kinetics were adjusted via subjectively obtained parameterizations by empirical observation of experienced clinicians (ENT) at nasofibroscopy. The dynamic MRI of swallowing will provide quantitative data on the velocities and amplitudes of the movements of the different anatomical structures present within SWALL-E: tongue base, epiglottis, pharyngeal constructor muscles, vocal cords and upper esophageal sphincter.

Transposing the data collected via MRI will allow to improve the accuracy and coordination of the kinetics of the synthetically reproduced movements.

Furthermore, by transposing the MRI data to SWALL-E, the investigators will be able to synchronize SWALL-E with data collected from any swallowing MRI performed in patients.

To improve SWALL-E, it will be necessary to exploit objective numerical data: speed and amplitude of movement of the anatomical structures of the pharyngo-larynx, measured by swallowing MRIs. These numerical data will make it possible to create a typical parameterization to obtain a functioning of the device as close as possible to a "normal" (healthy) pharyngolaryngeal set. Once the "normal swallowing" settings are achieved, it will be possible to mimic different types of "pathological swallowing".

The SWALL-E swallowing simulator (anatomical duct and simulation bench including such a duct) was the object of a national patent registration in 2017 (with a supplement in 2018), under the reference FR3071347A1, transferred to the University Hospitals of Strasbourg.

Swall-E is controlled by Lab-Viex software but the data acquired at imaging will be processed on a video tracking software (APREX track-R&D) to then be transposed to SWALL-E.

ELIGIBILITY:
Inclusion Criteria:

* Subject, male or female, between 18 and 60 years of age, affiliated to a social health insurance scheme (beneficiary or beneficiary's assistant)
* Subject able to understand the objectives and risks of the research and to give a dated and signed informed consent
* Subject has been informed of the results of the prior medical examination
* Healthy subject with no clinical swallowing disorders
* For a woman of childbearing age, negative urine pregnancy test at the inclusion visit

Exclusion Criteria:

* Subject with a contraindication to MRI: presence of non-removable ferromagnetic body, pacemaker, medication delivered by an implanted pump, ventricular bypass, history of epilepsy
* Subjects allergic to pineapple or latex
* Claustrophobic subject
* Subject suffering from swallowing disorders
* Subject with galactosemia
* Subject with dysphonia/dysphagia or inspiratory dyspnea on physical examination
* Subject with a history of cervico-facial surgery and/or radiotherapy
* Subject with a history of malignant or benign cervicofacial lesion
* Subject who has undergone intubation or endoscopy of the upper aerodigestive tract in the 3 months preceding the MRI
* Subject suffering from a degenerative neurological pathology
* Subject suffering from cardiac or respiratory insufficiency
* Subject in an exclusion period (as determined by a previous or current study)
* Unable to provide subject with informed information (subject in emergency situation, difficulty understanding subject)
* Pregnancy and/or breastfeeding
* Subject under court protection
* Subject under guardianship or curatorship

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
To Collect dynamic swallowing MRI imaging data from healthy volunteers | 1 hour
  to process to define the anatomical structures of interest

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'ORL Hôpital de Hautepierre, Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No